CLINICAL TRIAL: NCT01343953
Title: A Prospective Phase II Study to Evaluate Cord Blood Transplantation in Inherited or Acquired Severe Aplastic Anemia Refractory or in Relapse After Immunosuppressive Therapy
Brief Title: Cord Blood Transplantation in Severe Aplastic Anemia
Acronym: APCORD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P090201
Record Dates: First submitted 2011-04-27; First posted 2011-04-28 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Hereditary Diseases; Acquired Aplastic Anemia; Relapse; Absence of an HLA Identical Donor
Keywords: severe aplastic anemia; cord blood transplantation
MeSH Terms: conditions — Genetic Diseases, Inborn; Recurrence; Anemia, Aplastic | interventions — Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cord Blood Transplantation (Experimental)
  Interventions: Procedure: Cord Blood Transplantation

INTERVENTIONS:
Procedure: Cord Blood Transplantation — One or 2 cord blood units containing alone or both together more than 4x107 frozen nucleated cells/Kg with no more than 2 out of 6 HLA mismatches between them and with the patients for acquired Severe Aplastic Anemia

SUMMARY:
This is a Prospective Phase II Study to evaluate Cord Blood Transplantation in Inherited or Acquired Severe Aplastic Anemia Refractory or in Relapse after Immunosuppressive Therapy in the absence of an HLA identical donor;

DETAILED DESCRIPTION:
This is a Prospective Phase II Study to evaluate Cord Blood Transplantation in Inherited or Acquired Severe Aplastic Anemia Refractory or in Relapse after Immunosuppressive Therapy in the absence of an Human Leucocyte Antigen (HLA) identical donor; 26 patients will be recruited, according to a one step Fleming design

ELIGIBILITY:
Inclusion Criteria:

* Age: 3-55 years old
* inherited aplastic anemia (with severe aplastic anemia criteria) or acquired aplastic anemia in relapse or treatment failure after immunosuppressive therapy without clonal evolution
* Karnovsky Index >= 60%
* Informed consent

Exclusion Criteria:

* HLA identical donor

Ages: 3 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2011-05; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 year

SECONDARY OUTCOMES:
Graft versus host disease | 2 years
Infectious episodes | 1 year
treatment related mortality | 100 days
overall survival | 5 years
adverse events | 1 year
karnofsky scale | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Regis Peffault de la Tour, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- saint Louis, Paris, France

REFERENCES:
- [Derived] Peffault de Latour R, Chevret S, Jubert C, Sirvent A, Galambrun C, Ruggeri A, Gandemer V, Cornillon J, Rialland F, Dalle JH, Forcade E, Bruno B, Paillard C, Rorlich PS, Salmon A, Furst S, Sicre de Fontbrune F, Rubio MT, Bay JO, Mohty M, Larghero J, Gluckman E, Socie G; Francophone Society of Bone Marrow Transplantation and Cellular Therapy. Unrelated cord blood transplantation in patients with idiopathic refractory severe aplastic anemia: a nationwide phase 2 study. Blood. 2018 Aug 16;132(7):750-754. doi: 10.1182/blood-2018-01-829630. Epub 2018 May 14. PMID 29760162